CLINICAL TRIAL: NCT01097109
Title: The Effect of Somatic Dysfunction of the Pelvis, Sacrum and Lower Lumbar Spine on Weight Bearing
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Andrew kusienski, NSUCOM Sports Medicine Department Chair, Nova Southeastern University
Other Study IDs: 02171013Exp.
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Somatic Dysfunctions of Pelvis; Somatic Dysfunctions of Sacrum; Somatic Dysfunctions of Lower Lumbar Spine; Weight-Bearing
Keywords: Effect of Somatic Dysfunctions of Pelvis; Effect of Somatic Dysfunctions of Sacrum; Effect of Somatic Dysfunctions of Lower Lumbar Spine; Weight-Bearing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to determine if somatic dysfunctions of the pelvis, sacrum and lower lumbar spine have an effect on weight bearing. Our subjects are young, healthy subjects without recent soft tissue or osseous injury, a less than predetermined leg length discrepancy or OMM/chiropractic treatment. Their leg lengths will be measured; weight-bearing will be measured using a specialized scale and somatic dysfunctions diagnosed to determine if any correlation exists.

DETAILED DESCRIPTION:
Most sources claim that in individuals with leg length discrepancies, they tend to place more weight through the shorter lower extremity.1,2 Few cases state that the opposite is true.3 Many health care practitioners diagnose leg length discrepancies. Osteopathic physicians who practice with Osteopathic Manipulative Medicine (OMM) will also diagnose leg length discrepancies. They use testing to evaluate whether a leg length discrepancy is structural or functional. A structural leg length discrepancy is associated with shortening of bony structures.4 The structures affected can be due to congenital defects, which result in possible structural shortening of the tibia or femur, slipped capital femoral epiphyses (SCFE), or congenital dislocation. Other causes of structural leg length discrepancies include post total hip replacement, infections, tumors, paralysis, and trauma, including fractures where the gross length of a limb is altered.4 A structural leg length discrepancy can be most accurately assessed by physically measuring the distance between the anterior superior iliac spine (ASIS) and medial malleolus.4 The most reliable method of diagnosing a structural short leg is through full body radiographs. 6 A functional leg length discrepancy is a result of altered mechanics of the lower extremities. It is thought that a functional short leg occurs secondarily to a rotated pelvis caused by joint contractures and/or axial misalignments, including scoliosis.4 In osteopathic literature; functional leg length discrepancies are also thought to be the result of altered positions of the pelvis and sacrum. It is also thought in osteopathic philosophy that the position of the fifth lumbar vertebra affects the position of the sacrum. Therefore dysfunction of L5 will change the position of the sacrum such that a functional short leg is created.2(p.780-782) A common cause of functional leg length discrepancies diagnosed by osteopathic physicians is that of sacral base unleveling.5 The way in which a leg length discrepancy causes unleveling of the sacrum is through the femoral head of the longer leg driving the pelvis into a posterior rotation via forces placed through acetabular contact. Then the pelvis will typically rotate forward in attempts to lengthen the shorter leg, causing the sacral base to become unlevel.5 In addition, the sacral base tilts toward the side of the short leg.6 Standing postural x-rays, which outline sacral declination, are often used by chiropractors and osteopathic physicians to diagnose functional leg length discrepancies.6 Another way that functional leg length discrepancies are confirmed is through the supine to long sitting test, which tests for the presence of innominate rotations that may affect leg length as the cause.

There is no research known to support the presence of somatic dysfunctions, leg length discrepancies and altered weight bearing through lower extremities secondary to this.

It is common practice among osteopathic physicians who utilize OMM to diagnose musculoskeletal somatic dysfunctions of the pelvis, sacrum and lumbar spine. All these findings can contribute to low back pain. Therefore, it is the common practice of these physicians to diagnose leg length discrepancies, as it may ultimately result in low back pain.

Somatic dysfunction in osteopathic nomenclature is defined as 'impaired or altered function of related components of the somatic (body framework) system: Skeletal, arthrodial and Myofascial structures, and related vascular, lymphatic and neural elements'.2

There are specific somatic dysfunctions that lead to leg length differences. These effects include the sacral base tilting toward the side of the short leg, a low iliac crest on the short leg side, a forward rotation of the innominate on the shorter side and/or a posterior rotation of the innominate on the side of the longer leg as a compensatory measure. The lumbar spine will develop a convexity toward the side of the short leg.6 Their definitions are as follows:

Anteriorly rotated innominate: Entire innominate appears to be rotated anterior in relation to the opposite innominate. The ASIS will be more inferior or caudad and PSIS will be more superior or cephalad.2(776-778), 6 Posteriorly rotated innominate: Entire innominate appears to be rotated posterior in relation to the opposite hip bone. The ASIS will be more superior or cephalad and the PSIS more inferior or caudad.2(776-778), 6 Superior shear of the innominate: ASIS, PSIS and pubic ramus is more superior or cephalad than the opposite side.2(776-778), 6 Inferior shear of the innominate: ASIS, PSIS and pubic ramus is more inferior or caudad than the opposite side.2(776-778), 6

The way that osteopathic physicians determine the side of the somatic dysfunction is through the ASIS compression test. This is defined as follows:

ASIS compression test: Test for lateralization of somatic dysfunction of the sacrum, innominate or pubic symphysis. A posterior compression normally produces a palpatory sense of 'give' or 'resilience' as the innominate glides slightly posterior at the sacroiliac joint on that side. Somatic dysfunction of the pelvis on the side of compression produces resistance to the test determining the side of lateralization which is analogous to the determining the dysfunctional side. This is interpreted as a positive ASIS compression test.2(777) Individuals who have suffered from any type of osseous or soft tissue traumatic injuries in the last three months do not make suitable subjects for an evaluation of somatic dysfunctions' effects on weight bearing. Neither do individuals who have suffered from any type of osseous or soft tissue injuries in the lower extremity joints (knee, ankle, hip) in the last twelve months. As stated earlier, leg length discrepancies may be a result of trauma. Individuals who have suffered traumatic injuries within the last three months may exhibit antalgic or compensatory postures which may displace weight bearing more through one lower extremity than the other.7 This will ensure that the treatment population will be as homogenous as possible and will improve reliability of the study.

Individuals who have suffered lower extremity injuries in the last twelve months may also exhibit altered weight bearing distribution through the lower extremities. This may be something, depending on the chronicity of the problem, which alters weight bearing for an extended period of time which may vary depending on the person.7 Therefore, excluding individuals who have suffered lower extremity trauma in the last twelve months will also be excluded from the study to allow for more homogenous characteristics of our sample population. The time constraints of three and twelve months respectively were deemed as the exclusion times purely from anecdotal and clinical experience with lower extremity injury from the principal investigator and his colleagues.

1. White, S.C., Gilchrist, L.A., Wilk, B.E. Asymmetric limb loading with true or simulated leg-length differences. Clinical Orthopedics and Related Research, 2004,421,287-292
2. Ward, R. Foundations for Osteopathic Medicine 2nd Edition. 2003, p. 614-618, 780
3. McCaw, S.T., Bates, B.T. Biomechanical implications of mild leg length inequality. British Journal of Sports Medicine, 1991, 25,10-13
4. Gurney, B. Review: Leg length discrepancy. Gait and Posture. 2002, 15,195-206
5. Dott, G.A., Hart, C.L., McKay, C. Predictability of sacral base levelness based on iliac crest measurements. JAOA, 1994,4, 383-390.
6. DiGiovanna, EL. Schiowitz S. An Osteopathic Approach to Diagnosis and Treatment. Philadelphia: Lippincott-Raven, 301.
7. Riegger-Krugh, C & Keysor, J.J. Skeletal malalignments of the lower quarter: Correlated and compensatory motions and postures. J. Orthop Sports Phys Ther. 1996;23(2):164-170.

ELIGIBILITY:
Inclusion Criteria:

* Medical students of Nova Southeastern University College of Osteopathic Medicine (NSUCOM) ages 18-40.

Exclusion Criteria:

* individuals who have suffered from any type of osseous or soft tissue traumatic injuries in the last three months.
* individuals who have suffered from any type of osseous or soft tissue injuries in the lower extremity joints (knee, ankle, hip) in the last twelve months.
* anyone who has received either osteopathic or chiropractic manipulation within two weeks prior to taking part in the study.
* anyone who has a leg length difference of greater than one-quarter inch.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical students of Nova Southeastern University College of Osteopathic Medicine (NSUCOM) ages 18-40.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Kusienski, D.O., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University College of Osteopathic Medicine, Fort Lauderdale, Florida, United States

REFERENCES:
- [Background] White SC, Gilchrist LA, Wilk BE. Asymmetric limb loading with true or simulated leg-length differences. Clin Orthop Relat Res. 2004 Apr;(421):287-92. doi: 10.1097/01.blo.0000119460.33630.6d. PMID 15123962
- [Background] McCaw ST, Bates BT. Biomechanical implications of mild leg length inequality. Br J Sports Med. 1991 Mar;25(1):10-3. doi: 10.1136/bjsm.25.1.10. PMID 1913023
- [Background] Gurney B. Leg length discrepancy. Gait Posture. 2002 Apr;15(2):195-206. doi: 10.1016/s0966-6362(01)00148-5. PMID 11869914
- [Background] Dott GA, Hart CL, McKay C. Predictability of sacral base levelness based on iliac crest measurements. J Am Osteopath Assoc. 1994 May;94(5):383-90. PMID 8056627
- [Background] Riegger-Krugh C, Keysor JJ. Skeletal malalignments of the lower quarter: correlated and compensatory motions and postures. J Orthop Sports Phys Ther. 1996 Feb;23(2):164-70. doi: 10.2519/jospt.1996.23.2.164. PMID 8808518
- [Background] Ward, R. Foundations for Osteopathic Medicine 2nd Edition. 2003, p. 614-618, 780
- [Background] DiGiovanna, EL. Schiowitz S. An Osteopathic Approach to Diagnosis and Treatment. Philadelphia: Lippincott-Raven, 301.
- [Derived] Qureshi Y, Kusienski A, Bemski JL, Luksch JR, Knowles LG. Effects of somatic dysfunction on leg length and weight bearing. J Am Osteopath Assoc. 2014 Aug;114(8):620-30. doi: 10.7556/jaoa.2014.127. PMID 25082970